CLINICAL TRIAL: NCT03355118
Title: Exploring New Grounds in Physiology of the Elderly- Oxygen Extraction and Delivery During Anaesthesia and Major Surgery
Brief Title: Oxygen Extraction and Delivery in Elderly During Major Surgery
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Sigridur Kalman, Professor, Senior Consultant, Karolinska Institutet
Other Study IDs: K2017-0373; 4-500/2017 (Other: Karolinska Institutet)
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Impaired Oxygen Delivery; Surgery; Postoperative Complications; Peroperative Complication
MeSH Terms: conditions — Postoperative Complications; Intraoperative Complications | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: General anaesthesia and major surgery — The effect of general anaesthesia and surgery on oxygen transport and how it relates to outcome

SUMMARY:
This clinical observational study investigates perioperative oxygen consumption and delivery in elderly patients undergoing major surgery. The primary objectives are to characterise the perioperative oxygen delivery, consumption and potential markers of oxygen debt. Secondary objective is to estimate the correlation between oxygen delivery/consumption and postoperative outcomes to guide the design of a future trial.

DETAILED DESCRIPTION:
Background Intra- and postoperative fluid therapy aims to achieve or maintain pre-specified thresholds of oxygen delivery/blood flow which can be accomplished by use of fluids with or without inotropic drugs. The used thresholds of oxygen delivery were suggested over 40 years ago, in considerably younger patients compared to the current patients. Update of the characteristics of perioperative oxygen delivery and consumption is reasonable in modern clinical settings.

Primary outcome:

relative changes of oxygen consumption induced by anaesthesia

Secondary outcomes:

relative changes of oxygen consumption and delivery during surgery and postoperatively, oxygen extraction ratio (measured and estimated), potential markers of oxygen debt frequency of in-hospital postoperative complications, mortality (30 Days)

Population:

Men and women ≥65 years undergoing major/complex surgical procedures, when intra-operative cardiovascular monitoring is justified according to clinical decision.

Intervention: no study related intervention, general anaesthesia and surgery according to clinical routine

Blinding: no blinding

Study size:

Pilot study 1: feasibility assessment of study protocol of intra-operative measurements (n= max 10) Pilot study 2: feasibility assessment of study protocol of postoperative measurements (n= max 10) Main study: 60 subjects (20+´40) Planned analysis of oxygen consumption after 20 monitored subjects

Study duration:

Duration of haemodynamic monitoring 24-36 hours Duration of observation of clinical outcomes: 7-10 days, mortality at 30 days postop.

Investigational events:

monitoring of oxygen consumption and delivery monitoring of postoperative clinical outcomes monitoring of markers of tissue injury

Assessments, Procedures and Schedule of Investigational Events:

Subjects are identified by the operation planning list and assessed for eligibility. The study information will be given verbal during the first hospital visit. Subjects who give written informed consent will be included in the study.

Measurements:

oxygen consumption by indirect calorimetry via face mask (in awake state) and via expiratory extension tube of anaesthesia machine (unconscious state) cardiac output monitoring via arterial line (LiDCO) blood samples: arterial and venous blood gase samples, Troponin-T urine samples: N-gal

Clinical outcomes:

Data collection from medical records on postoperative complications using the POMS (postoperative morbidity survey) screening survey at days 3,7 and 10. Postoperative mortality at day 30.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged ≥65 years
2. Major/complex surgery (BUPA AXA classification of surgical severity)
3. Central and arterial venous catheterization for hemodynamic monitoring.
4. Written informed consent
5. Available research team for the measurements If two subjects are eligible the elder one will be chosen. If there are two subjects eligible of different gender and almost the same age, the subject with a gender that is underrepresented by two or more will be chosen. This is consistent with the purpose of including subjects with as high age as possible without interfering with recruitment.

Exclusion Criteria

1. Concomitant medication with Lithium (interferes with calibration of the LiDCO monitor)
2. Weight≤ 40 kg.
3. Not possible to establish arterial or central venous line.
4. Planned postoperative care at high-dependency unit (POP/IMA) <12hrs.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Men and women ≥65 years undergoing major/complex surgical procedures at the Karolinska University Hospital in Huddinge, Stockholm
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-04-04 (Actual)

PRIMARY OUTCOMES:
oxygen consumption | prior to and 15 minutes after anaesthesia induction
  change of oxygen consumption after anaesthesia induction

SECONDARY OUTCOMES:
oxygen consumption | perioperatively 0-36hrs
  changes of oxygen consumption during surgery and postoperative recovery
oxygen extraction ratio | perioperatively 0-36hrs
  ratio between oxygen consumption and oxygen delivery
oxygen extraction ratio: estimated and measured | perioperatively 0-36hrs
  ratio between oxygen consumption and oxygen delivery estimated from blood gases and measured by indirect calorimetry and cardiac output monitoring
C(v-a)pCO2/C(a-v)O2 | perioperatively 0-36hrs
  Ratio: venoarterial pCO2 difference/arterio-venous oxygen content difference
postoperative complications | postoperative days 3,5 and 10
  postoperative complications described by Postoperative Morbidity Survey (8)
mortality | postoperative days 30
  postoperative mortality

CONTACTS AND LOCATIONS:
Overall Officials: Erzsebet Bartha, MD PhD, Study Director — Karolinska University Hospital Huddinge, Stockholm, Sweden; Julia Jakobsson, MD, Principal Investigator — Karolinska University Hospital Huddinge, Stockholm, Sweden
Locations (1):
- Karolinska University hospital Huddinge, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jakobsson J, Noren C, Hagel E, Kalman S, Bartha E. Peri-operative oxygen consumption revisited: An observational study in elderly patients undergoing major abdominal surgery. Eur J Anaesthesiol. 2021 Jan;38(1):4-12. doi: 10.1097/EJA.0000000000001302. PMID 32858583